CLINICAL TRIAL: NCT01114178
Title: Estimation de la capacité Fonctionnelle à la Marche Par Questionnaire Clinique Chez Des Patients adressés Pour un Test de Marche Sur Tapis Roulant
Brief Title: Walking Impairment Questionnaire in PAD
Acronym: WELCH
Status: Terminated | Type: Observational
Why Stopped: recruitment problem due to administrative process being too long
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PL 2009/14
Record Dates: First submitted 2010-04-28; First posted 2010-05-03 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Peripheral Artery Disease
Keywords: questionnaire; peripheral artery disease; exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- claudicants: patients referred for a treadmill test
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — self completed questionnaire supervised by a technician

SUMMARY:
Purpose is to test and validate a new questionnaire (the WELCH questionnaire) to estimate walking capacity in patients with claudication

DETAILED DESCRIPTION:
Questionnaires (WELCH and WIQ) submitted to patients referred for treadmill walking test Comparison of sore to MWD on treadmill. Comparison with WIQ will be performed

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed, french language fluent patients

Exclusion Criteria:

* rejection of the questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients referred for treadmill testing
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
scoring of the WELCH questionnaire | 1 day
  predetermined score for the WELCH questionnaire answers (4 questions)

CONTACTS AND LOCATIONS:
Overall Officials: denise Jolivot, MD, Study Chair — University Hospital
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Fouasson-Chailloux A, Abraham P, Vielle B, Laporte I, Omarjee L, Ouedraogo N. The correlation of the "Walking Estimated-Limitation Calculated by History" (WELCH) questionnaire with treadmill maximal walking time is not impaired by age, in patients with claudication. Qual Life Res. 2015 Aug;24(8):1857-64. doi: 10.1007/s11136-015-0915-9. Epub 2015 Jan 13. PMID 25578404
- [Derived] Abraham P, Godet R, Harbonnier M, Laneelle D, Leftheriotis G, Ouedraogo N. External validation of the "walking estimated limitation calculated by history" (WELCH) questionnaire in patients with claudication. Eur J Vasc Endovasc Surg. 2014 Mar;47(3):319-25. doi: 10.1016/j.ejvs.2013.11.010. Epub 2013 Dec 3. PMID 24445082
- [Derived] Mahe G, Ouedraogo N, Marchand J, Vielle B, Picquet J, Leftheriotis G, Abraham P. Self-reported estimation of usual walking speed improves the performance of questionnaires estimating walking capacity in patients with vascular-type claudication. J Vasc Surg. 2011 Nov;54(5):1360-5. doi: 10.1016/j.jvs.2011.05.048. PMID 22027439
- [Derived] Mahe G, Ouedraogo N, Vasseur M, Faligant C, Saidi K, Leftheriotis G, Abraham P. Limitations of self-reported estimates of functional capacity using the Walking Impairment Questionnaire. Eur J Vasc Endovasc Surg. 2011 Jan;41(1):104-9. doi: 10.1016/j.ejvs.2010.10.002. Epub 2010 Nov 30. PMID 21123095